CLINICAL TRIAL: NCT04892420
Title: The Effect of Adding Dexamethasone Versus Magnesium Sulphate Versus Dexmedetomidine to Bupivacaine in Ultrasound Guided Adductor Canal Block for Post-operative Analgesia Following Anterior Cruciate Ligament Repair
Brief Title: Comparison Between Adjuvants Added to Bupivacaine in Adductor Canal Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ismail Mohammed, lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R 87/2021
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia
Keywords: dexamethasone,; magnesium sulphate; dexmedetomidine; adductor canal block; anterior cruciate ligament repair
MeSH Terms: interventions — Dexamethasone; Dexmedetomidine; Magnesium Sulfate; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: using computer generated codes and opaque sealed envelopes:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group DX (Active Comparator): The patients receive 20ml plain bupivacaine (0.5%) + 8 mg dexamethasone (2ml) in adductor canal block after spinal anesthesia
  Interventions: Drug: Dexamethasone
- Group DM (Active Comparator): The patients receive 20 ml plain bupivacaine(0.5%)+25 microgram dexmedetomidine( diluted in 2 ml normal saline) in adductor canal block after spinal anesthesia .
  Interventions: Drug: Dexmedetomidine
- Group M (Active Comparator): The patients receive 20 ml plain bupivacaine(0.5%)+200 milligram magnesium sulphate (2 ml of magnesium 10%) in adductor canal block after spinal anesthesia.
  Interventions: Drug: Magnesium sulfate
- Group C (Placebo Comparator): The patients receive 20ml plain bupivacaine (0.5%) + 2 ml of Normal saline in adductor canal block after spinal anesthesia.
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Dexamethasone — The patients receive 20ml plain bupivacaine (0.5%) + 8 mg dexamethasone (2ml) in adductor canal block after spinal anesthesia.
  Other Names: decadrone
  Arms: Group DX
Drug: Dexmedetomidine — The patients receive 20 ml plain bupivacaine(0.5)+25 microgram dexmedetomidine( diluted in 2 ml normal saline) in adductor canal block after spinal anesthesia .
  Other Names: precedex
  Arms: Group DM
Drug: Magnesium sulfate — The patients receive 20 ml plain bupivacaine(0.5)+200 milligram magnesium sulphate (2 ml of magnesium 10%) in adductor canal block after spinal anesthesia.
  Other Names: english salt
  Arms: Group M
Drug: Bupivacain — The patients receive 20ml plain bupivacaine (0.5%) + 2 ml of Normal saline in adductor canal block after spinal anesthesia.
  Other Names: marcain
  Arms: Group C

SUMMARY:
Adult patients undergoing anterior cruciate ligament repair under Spinal Anaesthesia will be randomly assigned into one of the following groups (The Four study groups will receive the standard treatment in the form of spinal anesthesia and adductor canal block), using computer generated codes and opaque sealed envelopes:

1. Group DX(DEXAMETHASONE): The patients receive 20ml plain bupivacaine (0.5%) + 8 mg dexamethasone (2ml) in adductor canal block after spinal anaetthesia.
2. Group DM (dexmedetomidine)The patients receive 20 ml plain bupivacaine(0.5)+25 microgram dexmedetomidine( diluted in 2 ml normal saline) in adductor canal block after spinal anaetthesia.
3. Group M (magnesium sulphate):The patients receive 20 ml plain bupivacaine(0.5)+200 milligram magnesium sulphate (2 ml of magnesium 10%) in adductor canal block after spinal anaetthesia.
4. Group C(CONTROL): The patients receive 20ml plain bupivacaine (0.5%) + 2 ml of Normal saline in adductor canal block after spinal anaetthesia.

DETAILED DESCRIPTION:
All patients will clinically be assessed and routine preoperative investigations will be done; CBC, Coagulation profile, liver function tests, kidney function tests, fasting blood sugar and ECG.

B. Intraoperative settings:

On arrival of the patients to the operative room, electrocardiography, non-invasive blood pressure, and pulse oximetry will be applied.

Baseline parameters such as systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), heart rate (HR), and oxygen saturation (SpO2) will be also recorded, All patients in this study will be positioned similarly during the entire surgical procedure and the whole procedures will be done by the same team.

Intravenous (IV) line will be inserted, and IV lactated Ringer will be started.

For all groups, spinal anaesthesia will be performed using spinal needle of 25-G under complete aseptic conditions All participants will receive spinal anaesthesia using hyperbaric 0.5% bupivacaine 20 mg and fentanyl 25 µg.

ACB will be done in the study at the end of surgery.

Specific equipment required: 22-gauge 100mm length, short-beveled regional block needle, skin antiseptic solution, sterile gloves, the portable ultrasound machine.

In Group DX:

The patients received 20ml plain bupivacaine (0.5%) + 8 mg dexamethasone (2ml) Position patient supine with knee slightly flexed and leg externally rotated

* Cleaning the area with Povidone-iodine 10% (Betadine), stand to the side of the patient to be blocked with the ultrasound machine on the opposite side and the screen facing, placing a high frequency ultrasound probe on the anterior aspect of the patient's thigh, approximately mid-point between the inguinal crease and medial condyle, Identifying the femur (usually at a depth of 3-5cm although variable) and move probe medially until the trapezoid/boat shaped Sartorius' muscle is visualized. The femoral artery lies just under this muscle within the adductor canal. Considering the saphenous nerve is almost always too small to be reliably imaged and the aim of the technique is therefore, to deposit local anesthetic under Sartorius and around the femoral artery (i.e. within the adductor canal).
* Optimizing image, adjusting depth, gain and frequency settings as required, the appropriate probe position is just proximal to where the femoral artery "dives" posteriorly and the probe should be positioned perpendicular to the artery. At this point the femoral artery should start to pass deeper to form the popliteal artery, the vastus medialis muscle lies anterolateral, the adductor magnus muscle posteromedial and the sartorius muscle medial. Use an in-plane approach from lateral to medial ensuring that your needle tip can be seen at all times, advance your needle into the adductor canal. This can be achieved by traversing Sartorius or Vastus Medialis, Aspirate and inject a test dose of 1 ml of the local anesthetic solution, observe the spread of the local anesthetic to ensure your needle tip is definitely within the adductor canal. If you cannot clearly see the spread of local anesthetic consider intravascular placement of needle and reposition, continue with the injection, aspirating every 5mls.

  2-In GROUP DM: 25 microgram dexmedetomidine will be Added.

  3-IN GROUP M: 200 milligram magnesium sulphate will be added

  4-IN GROUP C (CONTROL): Nothing will be added to bupivacaine.

C. Postoperative settings:

After the patient will be discharged from the operating room. Visual analog scale (VAS) will be used to assess the postoperative pain;

* The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a hand written mark on a 10-cm line that represents a continuum between "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm), and an eight-point verbal rating score for pain at rest (no pain _ 0, just noticeable _ 1, mild _ 2, weak _ 3, moderate _ 4, strong _ 5, severe _ 6,excruciating _ 7, same random word display shown to each patient).
* If VAS ≥ 3 postoperatively, IV increment of morphine will be given 0.1 mg per Kg not to be repeated every less than 3 hours ,The times of the first request for postoperative analgesia and the number of injections will be recorded. Any side effects will be recorded as hypotension (systolic arterial pressure <90 mmHg), arrhythmia, bradycardia (HR <60 beat/min), nausea or vomiting, or any other complications. Atropine 0.5 mg will be given in response to bradycardia, 20 ml per kg lactated Ringer will be given in response to hypotension.
* If local anaesthetic toxicity occurred, cardiovascular and respiratory support and 20% intralipid bolus of 100 ml over 2-3 min will be given.
* HR and MBP will be measured upon arrival to the PACU and after 30 min, then every hour if the patients remain in the PACU.
* In the surgical ward, vital signs (HR, SBP, MBP, DBP) as well as pain intensity will be assessed every 2 hours during the first 6 hours and then every 6 hours there for 24 hours postoperatively. All patients will receive ketorolac 30 mg IM every 8h. It will start immediately postoperatively in the PACU.

Measurements;

● Primary outcome:

VAS for pain (ranging from 0 to 10, where 0 no pain and 10 maximum pain) will be evaluated postoperatively and every 2 hours during the first 6 hours and then every 6 hours there for 24 hours postoperatively

Duration of postoperative analgesia (the time from recovery to the first given dose of morphine)

Number of patients needed rescue analgesia.

● Secondary outcome:

The total dose of morphine used postoperatively/patient (rescue analgesia) for 24 h.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years.
2. Sex: Both sexes.
3. Height 155-170 cm.
4. American Society of Anaesthesiologists (ASA) Physical Status Class-I and II.
5. Scheduled for anterior cruciate ligament under spinal anaesthesia.

Exclusion Criteria:

1. Declining to give written informed consent.
2. History of allergy to the medications used in the study.
3. Contraindications to regional anesthesia (including coagulopathy and local infection).
4. Psychiatric disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
rescue analgesia time | first 24 hours postoperatively
  time to first analgesic requirement

SECONDARY OUTCOMES:
rescue analgesia | 24 hours
  total dose of morphine needed postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ismail Mohammed Ibrahim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No